CLINICAL TRIAL: NCT06421142
Title: Application Research of FAPI Positron Emission Tomography(PET)/MRI, 18F-Fluorodeoxyglucose (FDG) PET/MRI, and MRI in the Diagnosis of Muscular Invasive Bladder Cancer and Evaluation of Neoadjuvant Therapy Efficacy
Brief Title: FAPI and FDG PET/MRI in Diagnosis and Therapy Prediction of Bladder Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ning Xu, Deputy Director of Department, First Affiliated Hospital of Fujian Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-041-02
Record Dates: First submitted 2024-05-09; First posted 2024-05-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-09

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Neoadjuvant Chemotherapy; Neoplasm Staging
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: In the MIBC diagnostic study and neoadjuvant efficacy prediction study, each patient underwent FAPIPET/MRI, FDGPET/MRI and MRI examinations, and were grouped and analyzed according to different examination methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- MIBC diagnostic study-FAPI PET/MRI (Experimental): suspected MIBC participants receive FAPI PET/MRI examination after entering the group.
  Interventions: Procedure: imaging examinations:FAPI PET/MRI, FDG PET/MRI, MRI
- MIBC diagnostic study-FDG PET/MRI (Experimental): suspected MIBC participants receive FDG PET/MRI examination after entering the group.
  Interventions: Procedure: imaging examinations:FAPI PET/MRI, FDG PET/MRI, MRI
- MIBC diagnostic study-MRI (Active Comparator): suspected MIBC participants receive MRI examination after entering the group.
  Interventions: Procedure: imaging examinations:FAPI PET/MRI, FDG PET/MRI, MRI
- MIBC neoadjuvant evaluation study-FAPI PET/MRI (Experimental): Patients diagnosed with MIBC receive FAPI PET/MRI examination before and after neoadjuvant therapy.
  Interventions: Procedure: imaging examinations:FAPI PET/MRI, FDG PET/MRI, MRI
- MIBC neoadjuvant evaluation study-FDG PET/MRI (Experimental): Patients diagnosed with MIBC receive FDG PET/MRI examination before and after neoadjuvant therapy.
  Interventions: Procedure: imaging examinations:FAPI PET/MRI, FDG PET/MRI, MRI
- MIBC neoadjuvant evaluation study-MRI (Active Comparator): Patients diagnosed with MIBC receive MRI examination before and after neoadjuvant therapy.
  Interventions: Procedure: imaging examinations:FAPI PET/MRI, FDG PET/MRI, MRI

INTERVENTIONS:
Procedure: imaging examinations:FAPI PET/MRI, FDG PET/MRI, MRI — FAPI PET/MRI and FDG PET/MRI examination Data acquisition was performed using a GE Healthcare SIGNA PET/MR instrument. Enrolled patients were injected intravenously with 68Ga-FAPI or 18F-FDG tracer and underwent simultaneous PET and MRI scanning approximately 30-60 minutes after intravenous administration of the tracer at a dose of 1.85-3.7 MBq/kg.
  MRI examination MRI examination was performed using a Skyra 3.0T MRI scanner from Siemens, Germany, with a 16-channel phased-array surface coil, and the scanning range was from the superior margin of the iliac wing to the inferior margin of the pubic symphysis.

SUMMARY:
The aim of this trial is to investigate the value of FAPI PET/MRI, FDG PET/MRI and MRI in diagnosing MIBC and predicting the efficacy of neoadjuvant therapy for MIBC patients, so as to guide the clinic to adjust the treatment plan in time and benefit MIBC patients.

DETAILED DESCRIPTION:
The MIBC diagnostic study was a prospective trial. According to the inclusion and exclusion criteria, patients with suspected MIBC were enrolled and underwent FAPI PET/MRI, FDG PET/MRI and MRI examination, and the imaging data and clinical laboratory and pathologic data were collected, and the postoperative pathological results were used as the gold standard to compare the accuracy of FAPI PET/MRI, FDG PET/MRI and MRI in diagnosing MIBC.

The MIBC neoadjuvant therapy efficacy assessment study was a prospective trial. Patients with MIBC were enrolled according to the inclusion and exclusion criteria, the regimen was selected individually according to the patient's condition, and the indicators were followed up until the end of time or the occurrence of an endpoint event to obtain information on survival time. FAPI PET/MRI, FDG PET/MRI and MRI were performed once before the start of neoadjuvant therapy and once after the end of therapy, and after the end of neoadjuvant therapy, patients received transurethral cystectomy of bladder tumors or radical cystectomy according to the efficacy and condition, and the combination of the imaging data and the clinical laboratory and pathological data were used to compare FAPI PET/MRI, FDG PET/ MRI and MRI in the assessment of the efficacy of neoadjuvant therapy in MIBC patients to guide clinical treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for MIBC diagnostic studies

  1. Patients with suspected muscle-invasive bladder cancer;
  2. Completion of FAPI PET/MRI, FDG PET/MRI and MRI;
  3. Complete clinical laboratory and pathological data.
* Inclusion criteria for MIBC neoadjuvant therapy efficacy evaluation study

  1. Patients diagnosed with muscle invasive bladder cancer;
  2. Completion of FAPI PET/MRI, FDG PET/MRI, and MRI before neoadjuvant therapy;
  3. Complete clinical laboratory and pathological data.

Exclusion Criteria:

* Exclusion criteria for MIBC diagnostic study

  1. Combined with other malignant tumors;
  2. Not receiving surgical treatment;
  3. Receiving neoadjuvant therapy before surgery;
  4. Previous allergy to contrast components or similar components;
  5. Serious organ function abnormalities, such as heart, lung, liver, kidney function serious abnormalities;
  6. Incomplete clinicopathological data
* Exclusion criteria of MIBC neoadjuvant therapy efficacy evaluation study

  1. Combination of other malignant tumors;
  2. FAPI PET/MRI, FDG PET/MRI and MRI were not completed after neoadjuvant therapy;
  3. Prior hypersensitivity to contrast components or similar components;
  4. Serious organ function abnormalities, such as serious abnormalities of heart, lung, liver and kidney function;
  5. Incomplete clinicopathological data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Sensitivity | Within 1 week after obtaining the surgical pathology report and imaging report results
  It is the percentage of patients who will be correctly judged as positive (true positive) if they actually have muscle invasive bladder cancer. The formula is TP/(TP+FN)×100%.TP is true positive and FN is false negative.
Diagnostic Specificity | Within 1 week after obtaining the surgical pathology report and imaging report results
  the percentage of patients who are not actually suffering from muscle invasive bladder cancer correctly judged as negative (true negative). The formula is TN/(TN+FP)×100%.TN is true negative, FP is false positive.
Positive Expected Value (PPV) | Within 1 week after obtaining the surgical pathology report and imaging report results
  the ratio of true positives among the positive results obtained by a specific test method. The formula is: PPV=TP/(TP+FP)×100%.
Negative Expected Value (NPV) | Within 1 week after obtaining the surgical pathology report and imaging report results
  refers to the ratio of true negatives among the negative results obtained by a specific test method. The formula is: NPV=TN/(TN+FN)×100%.
Positive Likelihood Ratio (PLR) | Within 1 week after obtaining the surgical pathology report and imaging report results
  the ratio of the probability that a patient who actually has muscle invasive bladder cancer is judged to be positive to the probability that a patient who actually does not have muscle invasive bladder cancer is judged to be positive. The formula was calculated as +LR = sensitivity/(1-specificity) × 100%.
Negative Likelihood Ratio (NLR) | Within 1 week after obtaining the surgical pathology report and imaging report results
  the ratio of the probability that a patient who actually has muscle invasive bladder cancer is judged negative to the probability that a patient who actually does not have muscle invasive bladder cancer is judged negative. The formula is: -LR=(1-sensitivity)/specificity×100%.
Youden Index | Within 1 week after obtaining the surgical pathology report and imaging report results
  the sum of sensitivity and specificity minus 1. Correct diagnostic index can be used for the comparison of two diagnostic methods, and the ideal correct diagnostic index is 100%. r = (specificity + sensitivity) - 1 = 1 - (false positive rate + false negative rate)
Standardized uptake values peak, maximum, and mean (SUVpeak , SUVmax, SUVmean) | Within 1 week after obtaining the surgical pathology report and imaging report results
  changes in SUVmax, SUVmean, and SUVpeak of the tumor lesion before and after treatment obtained from PET/MRI images.
Tumor-to-Background Ratio (TBR) | Within 1 week after obtaining the surgical pathology report and imaging report results
  changes in the ratio of the radioactivity of tumor tissue to the radioactivity of background tissue obtained from PET/MRI images before and after treatment.
Complete Remission (CR) | Within 1 month after obtaining the surgical pathology report and imaging report results
  In RECIST 1.1 Efficacy assessment criteria for conventional imaging, CR was defined as the disappearance of all target lesions, the absence of new lesions, and the normalization of tumor markers for at least 4 weeks. In PERCIST 1.1 efficacy evaluation criteria for FAPI PET/MRI and FDG PET/MRI, CR refers to the complete disappearance of tracer uptake.
Partial Remission (PR) | Within 1 month after obtaining the surgical pathology report and imaging report results
  In RECIST 1.1 Efficacy assessment criteria for conventional imaging, PR was defined as a decrease of ≥30% in the sum of the largest diameters of target lesions for at least 4 weeks. In PERCIST 1.1 efficacy evaluation criteria for FAPI PET/MRI and FDG PET/MRI, PR refers to a decrease of >30% in the peak SUV.
Stable Disease (SD) | Within 1 month after obtaining the surgical pathology report and imaging report results
  In RECIST 1.1 Efficacy assessment criteria for conventional imaging, SD was defined as a decrease in the sum of the largest diameters of the target lesions that did not reach PR or an increase in the size of the largest diameters of target lesions that did not reach PD. In PERCIST 1.1 efficacy evaluation criteria for FAPI PET/MRI and FDG PET/MRI, SD refers to a decrease of >30% in the peak SUV.
Progressive Disease (PR) | Within 1 month after obtaining the surgical pathology report and imaging report results
  In RECIST 1.1 Efficacy assessment criteria for conventional imaging, PD was defined as an increase in the sum of the largest diameters of the target lesions by at least ≥20% or the emergence of new lesions. In PERCIST 1.1 efficacy evaluation criteria for FAPI PET/MRI and FDG PET/MRI, PD refers to an increase of >30% in the peak SUL or the appearance of new lesions.
Complete Metabolic Response (CMR) | Within 1 month after obtaining the surgical pathology report and imaging report results
  For participants receiving FAPI PET/MRI and FDG PET/MRI, according to EORTC efficacy assessment criteria, CMR refers to the complete disappearance of tracer uptake.
Partial Metabolic Response (PMR) | Within 1 month after obtaining the surgical pathology report and imaging report results
  For participants receiving FAPI PET/MRI and FDG PET/MRI, according to EORTC efficacy assessment criteria, PMR refers to a reduction in SUV of ≥15%-25% after one cycle of treatment and a reduction in SUV of >25% after greater than one cycle of treatment.
Stable Metabolic Disease (SMD) | Within 1 month after obtaining the surgical pathology report and imaging report results
  For participants receiving FAPI PET/MRI and FDG PET/MRI, according to EORTC efficacy assessment criteria, SMD refers to an increase in SUV of <25% or a decrease of <15%, and tumor no significant increase in the extent of uptake (>20% increase in maximum diameter)
Progressive Metabolic Disease (PMD) | Within 1 month after obtaining the surgical pathology report and imaging report results
  For participants receiving FAPI PET/MRI and FDG PET/MRI, according to EORTC efficacy assessment criteria, PMD refers to an increase in SUV value of >25% and a significant increase in the extent of tumor uptake (increase in the largest diameter of >20%), or the appearance of new foci.
Pathologic Response | Within 1 month after obtaining the surgical pathology report and imaging report results
  According to pathological efficacy assessment criteria, Pathological Complete Remission(pCR) refers to no detectable tumor (pT0) or residual cancer confined to the original site (pTis) after treatment. According to pathological efficacy assessment criteria, A decrease in tumor stage from cT2 (Muscle-Invasive Bladder Cancer - MIBC) to non-muscle-invasive bladder cancer (NMIBC), including stages pT0, pTis, pTa, and pT1, indicates a treatment-sensitive tumor and is considered a good pathologic response. Conversely, if the tumor stage remains the same or increases, it is considered a poor pathologic response.

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 years to 3 years after receiving treatment
  the duration from the time a patient receives systemic therapy to the time of death from any cause.
Radiographic Progression Free Survival (rPFS) | 1 years to 3 years after receiving treatment
  the duration from the start of treatment to the occurrence of imaging progression or death due to any cause (whichever occurs first). Conventional imaging (RECIST 1.1 criteria), and FAPI PET/MRI (PERCIST 1.0 criteria) were used to assess the imaging progression of patients after receiving treatment, respectively.
Overall Remission Rate (Objective Response Rate, ORR) | Within 1 month after obtaining the surgical pathology report and imaging report results
  usually includes patient cases with CR+PR. Among them, conventional imaging was used to assess the proportion of patients meeting the criteria for CR or PR using the RECIST 1.1 criteria; FAPI PET/MRI was used to assess the proportion of patients meeting the criteria for CR or PR using the PERCIST 1.0 criteria;
Disease Control Rate (DCR) | Within 1 month after obtaining the surgical pathology report and imaging report results
  usually includes the proportion of patients with CR+PR+SD. Among them, conventional imaging uses RECIST 1.1 criteria to assess the proportion of patients meeting the criteria of CR or PR or SD; FAPI PET/MRI uses PERCIST 1.0 criteria to assess the proportion of patients meeting the criteria of CR or PR or SD.

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Yi Xue, Master, Study Chair — First Affiliated Hospital of Fujian Medical University
Locations (1):
- first hospital affiliated of Fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
We have chosen not to share the individual participant data (IPD) from this clinical study due to privacy and confidentiality concerns, as well as potential proprietary interests. Additionally, sharing IPD requires considerable resources for data de-identification and preparation, which may not be feasible within the scope of this study. However, we remain committed to transparency and will provide summary results and findings through appropriate channels, ensuring the dissemination of key insights while safeguarding participant privacy and confidentiality